CLINICAL TRIAL: NCT03658876
Title: Predictors of Response to Iron and Erythropoietin Stimulating Agents
Acronym: PRIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14HH1987
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Renal Failure Chronic; Anemia
Keywords: Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Injections; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EPO group (Active Comparator)
  Interventions: Drug: Epoetin Beta
- Iron group (Active Comparator)
  Interventions: Drug: Iron Sucrose Solution for Injection

INTERVENTIONS:
Drug: Iron Sucrose Solution for Injection — 200mg iron sucrose given on 5 successive haemodialysis sessions
  Arms: Iron group
Drug: Epoetin Beta — Uptitration of epoetin beta dose. Scale as follows (in units /session): 0-1000-2000-3000-4000-6000-8000-12000
  Other Names: Neorecormon
  Arms: EPO group

SUMMARY:
The purpose of the study is to identify predictors of treatment response. This involves collected baseline clinical parameters and bloods for biochemical parameters prior to administering the study treatment. A positive outcome following treatment was defined as an uptitration of haemoglobin by greater than 5g/l within 2 months. The study evaluated the participants response to treatment against the clinical and biochemical information collected prior to treatment being received.

ELIGIBILITY:
Inclusion Criteria:

* All prevalent haemodialysis patients, established for greater than 3 months

Exclusion Criteria:

Inability to consent Bone marrow disorder Transfusion dependence Active bleeding Active infection Active malignancy Frail with either frequent hospital admissions or unable to follow trial protocol due to differing target haemoglobin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damien Ashby, MBBS, Principal Investigator — Imperial College Healthcare NHS Trust

IPD SHARING:
Plan to Share IPD: No
No indication to do so

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 197 individuals who consented to the study. These were in the observational phase. There were 184 randomisation episodes from these individuals.
Period: Overall Study
Arm/Group | Iron Group | EPO Group
Started | 88 | 96
Completed | 76 | 84
Not Completed | 12 | 12
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 0 | 1
Not completed — Intercurrent illness | 6 | 4
Not completed — Transplantation/other operation | 1 | 5

BASELINE CHARACTERISTICS:
Population: This study was analysed on a per protocol rather than intention to treat basis
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Group | EPO Group | Total
Number analyzed (Participants) | 76 | 84 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 41 | 78
  >=65 years | 39 | 43 | 82
Age, Continuous [Mean (Full Range); unit: years] | 63.22 [31 to 86] | 63.1 [25 to 91] | 63.16 [25 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 54 | 60 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 41 | 75
  Black | 9 | 12 | 21
  Asian | 31 | 28 | 59
  Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 76 | 84 | 160

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Incrementation
Description: Incrementation of haemoglobin of 5g/l following treatment
Time Frame: Within 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | EPO Group | Iron Group
Number analyzed (Participants) | 84 | 76
Participants | 61 | 53

ADVERSE EVENTS:
Arm/Group | Iron Group | EPO Group
All-Cause Mortality (participants affected / at risk) | 3/88 | 2/96
Serious Adverse Events (participants affected / at risk) | 17/88 | 21/96
Other Adverse Events (participants affected / at risk) | 2/88 | 1/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Group (N=88) | EPO Group (N=96)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 2 (2) — 1 episode of arrhythmia on dialysiand and one episode of atrial fibrillation with fast ventricular rate
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Soft tissue infection (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — 1 diabetic foot and 1 cellulitis
Cervical discitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1) — Hospital admission due to clinical concern of cardiac event
Vasculitis (Immune system disorders) | 0 (0) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — Following falls
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infection related to catheters (Infections and infestations) | 1 (1) | 1 (1) — Infections related to tunnelled haemodialysis access
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Psoas abscess (Infections and infestations) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Group (N=88) | EPO Group (N=96)
Transfusion (Blood and lymphatic system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No